CLINICAL TRIAL: NCT01994668
Title: A Phase 1, Randomized Single-blind (Subject-blind), Placebo Controlled Study to Characterize the Safety and Pharmacokinetics of Single Intravenous Dose of Lorazepam in Healthy Japanese Adult Subjects
Brief Title: Phase 1 Study to Characterize the Safety and Pharmacokinetics of Single Intravenous Dose of Lorazepam in Healthy Japanese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B3541001
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: lorazepam; intravenous; pharmacolinetics; healthy; Japanese
MeSH Terms: interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lorazepam (Experimental)
  Interventions: Drug: Lorazepam
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorazepam — A single intravenous administration of 2 mg lorazepam over 1 minute
  Arms: Lorazepam
Drug: Placebo — A single intravenous administration of 0.9% saline over 1 minute
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of 2-mg lorazepam intravenous administration in healthy Japanese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and/or female subjects of non-childbearing potential.
* Body Mass Index of 17.5 to 30.5 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

* History of sensitivity to lorazepam or other benzodiazepines.
* Evidence or history of acute narrow-angle glaucoma or sleep apnea syndrome.
* Significant psychiatric disorder, recurrent episodes of severe depression, or subjects with serious suicidal risk.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs). | Day 1 to Day 4
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1
Area under the Concentration-Time Curve (AUC) | Day1 to Day 4
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3541001&StudyName=Phase%201%20Study%20to%20Characterize%20the%20Safety%20and%20Pharmacokinetics%20of%20Single%20Intravenous%20Dose%20of%20Lorazepam%20in%20Healthy%20Japanese%20Adult%20Subjects